CLINICAL TRIAL: NCT07140003
Title: Microbiological Value of Sonographic Guided Pleural Tissue Culture Plus Pleural Fluid Culture in Patients With Infected Pleural Fluid
Brief Title: Pleural Tissue Culture Versus Pleural Fluid Culture in Infected Effusion
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: pleura,tissue culture,sonograp
Record Dates: First submitted 2025-08-12; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-07

CONDITIONS: Pleural Tissue Culture
Keywords: pleural tissue culture ,infected pleural fluid

STUDY DESIGN:
Intervention Model Description: MICROBIOLOGICAL VALUE OF SONOGRAPHIC GUIDED PLEURAL TISSUE CULTURE PLUS PLEURAL FLUID CULTURE IN PATIENTS WITH INFECTED PLEURAL FLUID
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- one group of patients will undergo pleural fluid culture taken by ultrasound chest by 18 gauge needl (Active Comparator): microbiological culture of the fluid
  Interventions: Procedure: pleural biopsy
- sonographic guided pleural tissue culture (Active Comparator): pareital pleural biobsy will be taken from the posterior costal pleura by ultrasound via true cut biopsy 12 french and tissue will be sent to the micro alab
  Interventions: Procedure: pleural biopsy

INTERVENTIONS:
Procedure: pleural biopsy — To assess whether pleural tissue culture can improve the identification of causative organisms in pleural infections (using the pleural fluid culture), which can aid in selecting appropriate antimicrobial therapy and improve treatment outcomes, thus may provide valuable insights into the utility of pleural tissue culture in managing pleural infection and may guide clinicians in selecting the most appropriate diagnostic approach.

SUMMARY:
comparison between the result of fluid culture and that of pleural tissue culture

DETAILED DESCRIPTION:
MICROBIOLOGICAL VALUE OF SONOGRAPHIC GUIDED PLEURAL TISSUE CULTURE PLUS PLEURAL FLUID CULTURE IN PATIENTS WITH INFECTED PLEURAL FLUID

ELIGIBILITY:
Inclusion Criteria:

* Exudate neutrophilic pleural fluid aspirate, or met at least one or more of the following criteria: grossly frank purulent, gram stain positive for bacteria, bacterial culture positive, acidic with a pH <7.20, low pleural fluid glucose (<55mg/dL), and CT evidence of pleural infection. Exclusion criteria: Pleural infections by Mycobacterium tuberculosis.Malignant effusion.Coagulation defects.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
initial pleural fluid and parietal pleural tissue | 2 weeks
  the result of culture
result of culture | one month
  the result of pleural fluid culture and the pleural tissue culture result

CONTACTS AND LOCATIONS:
Overall Officials: mohamed sabry eltarhony, lecturer, Principal Investigator — Alexandria University; hatem essam hamed, lecturer, Study Director — Alexandria University
Locations (1):
- Chest Department -Faculty of Medicine, Alexandria, Chest Department, Egypt

IPD SHARING:
Plan to Share IPD: No
according to the policy of ethics committee

REFERENCES:
- See also: national library of information — https://pubmed.ncbi.nlm.nih.gov/21793988/